CLINICAL TRIAL: NCT05653739
Title: Mindfulness Based Stress Reduction Intervention
Acronym: MBSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Irum Mir, PhD Scholar /Principle Investigator, Fatima Jinnah Women University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FJWU/EC/2022/46
Record Dates: First submitted 2022-11-19; First posted 2022-12-16 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Intervention Study

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Intervention Group (Experimental): Mindfulness Based Stress Reduction Intervention , The training consists of eight weekly group sessions with the duration of approximately 2-2.5 hours with a trained instructor. Further participants were given daily audio-guided home practice (approximately 45 min/day), and a day-long mindfulness retreat (occurring during week sixth of the 8-week program)
  Interventions: Behavioral: Mindfulness Based Stress Reduction Intervention
- Control Group (No Intervention): Participants in the control group were not given any intervention in order to compare with the experimental group. At the end of the study participants in this group were also offered relaxation trainings in order to deal with the psychological distress, quality of life and distress tolerance.

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction Intervention — MBSR is Mindfulness based intervention designed by Kabat-Zinn (1990) in order to deal with the stress and other psychological issues among individuals. This has been very effective intervention across different cultures . In this 8 week intervention participants will be given some home tasks to practice for at least 40 minutes a day.
  Arms: Mindfulness Based Intervention Group

SUMMARY:
The aim of the current study is to find out the impact of Mindfulness based stress reduction intervention on psychosocial factors associated with distress tolerance and quality of life among youth . The study is conducted on the youth age ranging from 15-24 years from districts Mardan and Nowshera of KP. Standardized tools are used to screen highly vulnerable cohort for further intervention. Eligible participants who scored higher on psychological distress, vicarious traumatization, and low on distress tolerance and quality of life and show their consent were recruited for the Intervention Phase. Participants were assigned randomly to experimental and control groups in intervention phase. Participants in the experimental group were given Mindfulness Based Stress Intervention (MBSR) training in the settings conducive for research.

ELIGIBILITY:
Inclusion Criteria:

* The participants studying in different public and private sector higher education institutes of Mardan and Nowshera districts of KP.
* Participants who volunteer to participate were included.
* Participants with High psychological distress, and Vicarious Trauma.
* Participants with low distress tolerance and low quality of life.

Exclusion Criteria:

* Participants below 15 years or above 24 years i.e., the age range of youth (as recommended by WHO) will be excluded.
* Participants with any significant reported medical disease were also excluded.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in Psychological distress. | Psychological distress will be measured before giving the intervention and at 8 weeks of intervention again the scale will be administered to measure psychological distress in order to check changes.
  Psychological distress will be measured through Depression Anxiety and Stress Scale (DASS). After giving intervention to the participants it is expected that the participants will score low on the scale as low score is the indication of low level of psychological distress on DASS. Score above 32 will be considered as high level of psychological distress while score below 32 will be considered as indication of low level of psychological distress
Changes in Vicarious Trauma | The time frame for the completion of intervention is 8 weeks after which it is expected that participants will score low on STQ.
  Vicarious Trauma will be measured through Secondary Stress Trauma Questionnaire. Individuals scoring above 44 on the scale is the indication of high level of secondary traumatic symptoms.
Change in Distress Tolerance | The time frame for the completion of intervention is 8 weeks after which it is expected that participants will score low on DTS i.e., their distress tolerance will be improved.
  Distress Tolerance will be measured through Distress Tolerance Scale (DTS).Low scores on the scale is the indication of higher level of distress tolerance. So score above 34 will be selected for participants to be recruited for study.
change in Quality of Life | The time frame for the completion of intervention is 8 weeks after which it is expected that participants will score high on WHOQOL-BREF.
  Quality of life will be measured through The World Health Organization Quality of Life Scale (WHOQOL-BREF). High scores on the scale is the indication of high level of quality of life. Individuals scoring above 62 on the scale will be considered as scoring high on QOL for the current study. After participants are exposed to the intervention they will score higher on WHOQOL-BREF which means high quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatima Jinnah Women University, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The findings of the study will be shared with the other researchers in the field through published research articles.

REFERENCES:
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Denollet J. DS14: standard assessment of negative affectivity, social inhibition, and Type D personality. Psychosom Med. 2005 Jan-Feb;67(1):89-97. doi: 10.1097/01.psy.0000149256.81953.49. PMID 15673629
- [Background] Motta RW, Kefer JM, Hertz MD, Hafeez S. Initial evaluation of the Secondary Trauma Questionnaire. Psychol Rep. 1999 Dec;85(3 Pt 1):997-1002. doi: 10.2466/pr0.1999.85.3.997. PMID 10672764
- [Background] Simons,J.S., Gaher,R.M.(2005). The Distress Tolerance Scale: Development and Validation of a Self Report Measure. Motivation and Emotion,29,83-102. https://doi.org/10.1007/s11031-005-7955-3
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712